CLINICAL TRIAL: NCT06419686
Title: The Separate and Combined Glucagonotropic Effects of Glucose-dependent Insulinotropic Polypeptide and Alanine in Healthy Individuals
Brief Title: The Glucagonotropic Effects of Glucose-dependent Insulinotropic Polypeptide and Alanine in Healthy Individuals
Acronym: GIPALANIN
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, MD PhD, Professor, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-21066812
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Effect of iv Administration of GIP and Alanine
MeSH Terms: interventions — Sodium Chloride; Alanine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Saline (Placebo Comparator): Intravenous administration of saline for 90 minutes.
  Interventions: Other: Placebo (saline)
- GIP (Experimental): Intravenous administration of GIP for 90 minutes (priming dose 6 pmol/kg/min for 10 minutes and 4 pmol/kg for 80 minutes.
  Interventions: Drug: GIP
- Alanine (Experimental): Intravenous administration of alanine for 90 minutes (28 umol/kg/min).
  Interventions: Drug: Alanine
- GIP + Alanine (Experimental): Intravenous administration of GIP and alanine for 90 minutes. GIP is given at a priming dose of 6 pmol/kg/min for 10 minutes and then 4 pmol/kg for 80 minutes. Alanine is given at 28 umol/kg/min for 90 minutes.
  Interventions: Drug: GIP + alanine

INTERVENTIONS:
Other: Placebo (saline) — Intravenous saline during experimental days.
  Arms: Saline
Drug: GIP — Intravenous GIP administration during experimental days.
  Arms: GIP
Drug: Alanine — Intravenous alanine administration during experimental days.
  Arms: Alanine
Drug: GIP + alanine — Intravenous administration of GIP and alanine during experimental days.
  Arms: GIP + Alanine

SUMMARY:
The study is a randomised, double-blinded, placebo-controlled, crossover study enrolling 10 healthy male participants. Each participant will undergo four separate study days in randomised order. Each study day encompasses a continous 90-minute i.v. infusion with either placebo, glucose-dependent insulinotropic polypeptide (GIP), alanine or GIP + alanine.

The primary objective of the study is to find out whether intravenous administration of the naturally occuring gut hormone GIP and the amino acid alanine, separately and combined, results in additive or synergistic glucagonotropic effects during euglycaemic conditions in healthy participants. Secondary objectives are to disclose the effect of the abovementioned interventions on insulin secretion and circulating levels of total and individual amino acids.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian ethnicity
* Body mass index (BMI) 20-27 kg/m^2
* Glycated haemoglobin (HbA1c) ≤ 42 mmol/mol
* Informed and written consent

Exclusion Criteria:

* Late microvascular complications except mild nonproliferative retinopathy
* Liver disease (alanine aminotransferase (ALAT) and/or aspartate aminotransferase (ASAT) > 2 times normal values) or history of hepatobiliary disorder
* Treatment with any glucose-lowering drugs
* Active or recent (within 5 years) malignant disease
* Active tobacco smoking/use
* Any condition considered incompatible with participation by the investigators.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Plasma concentrations of Glucagon | Timepoint -30 to 90 minutes
  Baseline
Plasma concentrations of Glucagon | Timepoint -30 to 90 minutes
  Baseline-corrected area under the curve (bsAUC)

SECONDARY OUTCOMES:
Serum concentration of Insulin | Timepoint -30 to 90 minutes
  Baseline
Serum concentration of Insulin | Timepoint -30 to 90 minutes
  Baseline-corrected area under the curve (bsAUC).
Serum concentration of C-peptid | Timepoint -30 to 90 minutes
  Baseline
Serum concentration of C-peptid | Timepoint -30 to 90 minutes
  Baseline-corrected area under the curve (bsAUC).
Plasma concentration of glucose | Timepoint -30 to 90 minutes
  Baseline
Plasma concentration of glucose | Timepoint -30 to 90 minutes
  Baseline-corrected area under the curve (bsAUC).
Plasma concentration of glucose | Timepoint -30 to 90 minutes
  Peak value
Plasma concentration of GIP | Timepoint -30 to 90 minutes
  Baseline
Plasma concentration of GIP | Timepoint -30 to 90 minutes
  Baseline-corrected area under the curve (bsAUC).
Circulating levels of total amino acids | Timepoint -30 to 90 minutes
  Baseline
Circulating levels of total amino acids | Timepoint -30 to 90 minutes
  Baseline-corrected area under the curve (bsAUC).
Circulating levels of individual amino acids | Timepoint -30 to 90 minutes
  Baseline
Circulating levels of individual amino acids | Timepoint -30 to 90 minutes
  Baseline-corrected area under the curve (bsAUC).
Lipid profile | Timepoint -30 to 90 minutes
  Baseline
Lipid profile | Timepoint -30 to 90 minutes
  Baseline-corrected area under the curve (bsAUC).
Circulating levels of CTx | Timepoint -30 to 90 minutes
  Baseline
Circulating levels of CTx | Timepoint -30 to 90 minutes
  Baseline-corrected area under the curve (bsAUC).
Circulating levels of P1NP | Timepoint -30 to 90 minutes
  Baseline
Circulating levels of P1NP | Timepoint -30 to 90 minutes
  Baseline-corrected area under the curve (bsAUC).
Blood pressure | Timepoint -30, 0, 30, 60, 90
  Baseline
Blood pressure | Timepoint -30, 0, 30, 60, 90
  Baseline-corrected area under the curve (bsAUC).
Pulse | Timepoint -30, 0, 30, 60, 90
  Baseline
Pulse | Timepoint -30, 0, 30, 60, 90
  Baseline-corrected area under the curve (bsAUC).

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD, PhD, Principal Investigator — Center for Clinical Metabolic Research, Gentofte Hospital
Locations (1):
- Center for Clinical Metabolic Research, Gentofte Hospital, Hellerup, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No